CLINICAL TRIAL: NCT01745874
Title: Diagnostic Value of Whole-Body MRI Compared to FDG-PET-CT for Rectal Cancer Preoperative Staging, Before and After Neoadjuvant Treatment
Brief Title: Diagnostic Value of Whole-Body MRI for Rectal Cancer Preoperative Staging
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Lausanne Hospitals (Other)
Responsible Party: Principal Investigator, Milena Cerny, Dr. Milena Cerny, University of Lausanne Hospitals
Other Study IDs: 247/12
Record Dates: First submitted 2012-12-02; First posted 2012-12-10 (Estimated); Last update posted 2012-12-10 (Estimated); Status verified 2012-12

CONDITIONS: Rectal Cancer
Keywords: Rectal cancer; Whole-body MRI; FDG-PET-CT; preoperative staging
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to determine whether whole-body MRI (WB-MRI) accuracy is superior to FDG-PET-CT considered as the gold-standard for the staging of distant lesions of rectal cancer.

DETAILED DESCRIPTION:
Rectal cancer is the second cause of mortality after lung cancer in industrialized countries and represent 28% of colorectal carcinomas. Despite major improvements in diagnosis and treatment made those last years,mortality and morbidity remains high, because of high prevalence of metastasis and local recurrence. A accurate initial staging is of paramount importance for an appropriate treatment (neoadjuvant chemiotherapy and radiotherapy, surgery).

Actually, there is no international consensus concerning imaging for the staging of rectal cancer and modalities used are variable from one center to another.

WB-MRI represented a attractive and promising technique for the staging of rectal cancer, free of ionizing radiation .

ELIGIBILITY:
Inclusion Criteria:

* rectal cancer T3 N+ or T3 or T4

Exclusion Criteria:

* renal failure
* allergy to iodinated contrast medium
* contraindication to MRI

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with a rectal cancer
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2012-10; Primary Completion 2013-10 (Estimated); Study Completion 2013-10 (Estimated)

PRIMARY OUTCOMES:
Evaluate the diagnostic accuracy of whole-body MRI for the staging of rectal cancer before and after neoadjuvant treatment | baseline and 1 week before surgery
  We will compare for each body region the findings of the whole-body MRI to the FDG-PET-CT considered as the gold-standard and measure sensibility/specificity and diagnostic accuracy of the whole-body MRI for distant lesions of rectal cancer.

SECONDARY OUTCOMES:
Tumoral regression after neoadjuvant treatment | baseline and six weeks after the end of the neoadjuvant treatment
  Evaluate the tumoral regression after neoadjuvant treatment on the MRI by the measurement of the ADC (attenuation diffusion coefficient) increase and compare the results to the measure of the SUV (standard uptake value) decrease on the FDG-PET-CT.

CONTACTS AND LOCATIONS:
Overall Officials: Milena Cerny, Principal Investigator — University of Lausanne Hospitals; Sabine Schmidt Kobbe, Dr., Principal Investigator — University of Lausanne Hospitals
Locations (1):
- University of Lausanne Hospitals, Lausanne, Canton of Vaud, Switzerland